CLINICAL TRIAL: NCT00002810
Title: Autologous Peripheral Blood Stem Cell Transplantation With High Dose Melphalan For Treatment Of Primary Amyloidosis (AL)
Brief Title: High-Dose Melphalan Followed by Peripheral Stem Cell Transplant in Treating Patients With Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Bone marrow Transplant Program, Temple University Health Systems
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000064938; TUHSC-2797; NCI-V96-0951
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; primary systemic amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Immunoglobulin Light-chain Amyloidosis | interventions — Filgrastim; Melphalan; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: melphalan
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of plasma cells, either by killing the cells or by stopping them from dividing. Having a peripheral stem cell transplant to replace the blood-forming cells destroyed by chemotherapy, allows higher doses of chemotherapy to be given so that more plasma cells are killed. By reducing the number of plasma cells, the disease may progress more slowly.

PURPOSE: This phase II trial is studying how well giving high-dose melphalan together with peripheral stem cell transplant works in treating patients with primary amyloidosis or amyloidosis associated with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess overall and progression-free survival following high-dose melphalan and autologous peripheral blood stem cell transplantation in patients with primary amyloidosis.
* Evaluate the toxic effects associated with this treatment regimen.
* Evaluate the function of involved organs, especially the heart, lungs, and nervous system, before and after treatment with this regimen.

OUTLINE: Peripheral blood stem cells (PBSC) are mobilized with granulocyte colony-stimulating factor (G-CSF) for 5 days and then collected by leukapheresis. Patients receive high-dose melphalan on 2 consecutive days, followed by 1 day of rest, then by PBSC transplantation. G-CSF is given from 1 day after transplantation until the neutrophil count is greater than 1,500 for 3 consecutive days.

Patients are followed at 100 days and 1 year post-transplant.

PROJECTED ACCRUAL: A very small number of patients are expected to be accrued over 5-10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Primary amyloidosis diagnosed by appropriate amyloid stains or electromicroscopy of abdominal fat, bone marrow, or other target tissues

  * Pathology reviewed by Temple University
* Amyloidosis secondary to any stage of multiple myeloma allowed provided plasma cell concentration in bone marrow is less than 15%
* No amyloidosis secondary to rheumatoid arthritis or chronic infection
* No familial amyloidosis

PATIENT CHARACTERISTICS:

Age:

* 16 to 65

Performance status:

* Karnofsky 80-100%

Hematopoietic:

* Not specified

Hepatic:

* Liver function tests less than twice normal
* No active liver disease

Renal:

* Creatinine clearance greater than 50 mL/min
* Nephrotic syndrome allowed

Cardiovascular:

* Cardiac evaluation required in patients with left ventricular ejection fraction less than 45% by echocardiogram or MUGA
* No poorly controlled hypertension

Pulmonary:

* FEV_1 and DLCO greater than 50% of predicted, or pulmonary evaluation required
* No chronic obstructive pulmonary disease

Other:

* No history of serious coagulopathy, hemorrhage, or bleeding
* No active infection
* No other serious comorbid disease (e.g., poorly controlled diabetes)
* No pregnant women
* Adequate contraception required of fertile women

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* More than 12 monthly cycles of prior alkylating agent chemotherapy discouraged

Endocrine therapy:

* Corticosteroids discontinued at least 6 weeks prior to transplantation

Radiotherapy:

* No prior radiotherapy

Surgery:

* Not specified

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-05; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Overall survival
Time to clinical progression of amyloid symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth F. Mangan, MD, FACP, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase-Temple Cancer Center CCOP Research Base, Philadelphia, Pennsylvania, United States